CLINICAL TRIAL: NCT06389630
Title: Evaluation of the Efficiency of Two Different Teaching Methods in Safe Subcutaneous Injection Skills in Type 2 Diabetes Mellitus Patients
Brief Title: Evaluation of the Efficiency of Two Different Teaching Methods in Safe Subcutaneous Injection Skills
Acronym: EETDTMSSİS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Sağlık ve Teknoloji Üniversitesi (Other)
Responsible Party: Principal Investigator, Azzet Yüksel, Lecturer,Principal Investigator, Kocaeli Sağlık ve Teknoloji Üniversitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0012
Record Dates: First submitted 2024-03-08; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-03

CONDITIONS: Complication of Injection
Keywords: video-assisted training; practice skill; nursing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video-assisted training group (Experimental)
  Interventions: Other: video-assisted training group
- low fidelity simulation model group (Experimental)
  Interventions: Other: low fidelity simulation model group

INTERVENTIONS:
Other: video-assisted training group — This group will be taught subcutaneous insulin injection through video-supported training.
  Arms: video-assisted training group
Other: low fidelity simulation model group — This group will be taught subcutaneous insulin injection on a low-fidelity simulation model.
  Arms: low fidelity simulation model group

SUMMARY:
Subject: Subcutaneous (SC) insulin injection is frequently used in the treatment of Type 2 Diabetes patients. Complications such as pain, ecchymosis, hematoma, lipoatrophy and lipohypertrophy are frequently observed after SC injections. These complications that develop due to incorrect injection application negatively affect the use of injection application areas, change body image and negatively affect drug absorption. In order to reduce and prevent complications related to SC insulin injection, it is very important to gain the skill of safe SC insulin injection. It is stated that there are a limited number of studies on which of the teaching methods used in sick individuals are effective. In the national and international literature, no study has been found evaluating the effect of SC injection skill teaching based on video-supported training and low-fidelity simulation model applications on disease management in individuals diagnosed with Type 2 Diabetes Mellitus. In this regard, the research was planned as an experimental design in order to examine the effectiveness of video-supported training and low-fidelity simulation model-based teaching in gaining safe insulin injection skills via SC. For this purpose; It is aimed to evaluate the effect of two different skill teaching methods on the patient's SC injection ability, complication management and blood glucose level.

Purpose: This research was planned as an experimental design to examine the effectiveness of two different teaching methods (video-supported training and low-fidelity simulation model) in gaining safe insulin injection skills via the Subcutaneous (SC) route.

Design: A pretest-posttest two-group, quasi-experimental design will be used in the study.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 years of age or older,
* Have the physical and mental ability to accurately evaluate the Visual Analog Scale (VAS),
* The platelet count is 100 000/mm3 and above,
* Having a diagnosis of Type 2 Diabetes Mellitus,
* No dementia according to Mini-Cog test evaluation,
* The plan was to agree to participate in the study.

Exclusion Criteria:

* Having verbal and auditory problems,
* Using oral or SC anticoagulant
* Presence of any findings such as scarring, incision, ecchymosis, hematoma, lipoarthrrophy and lipohypertrophy on the skin in the area where the injection will be made,
* Recurrent use of drugs that affect the formation of lipoatrophy and lipohypertrophy, such as octroid, corticosteroid, and antiretroviral therapy,
* It was defined as having a diagnosis of Diabetes during pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-04-29 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
subcutaneous injection skills | After 1 week, After 1 month, After 3 months
  The "subcutaneous injection checklist" will be used to measure patients' ability to administer subcutaneous injection.
ecchymosis | After 1 week, After 1 month, After 3 months
  "Opsite-Flexigrid Measurement Tool" will be used to measure ecchymosis that occur after subcutaneous injection.
hematoma | After 1 week, After 1 month, After 3 months
  Opsite-Flexigrid Measurement Tool" will be used to measure hematoma that occur after subcutaneous injection.
lipoarthrrophy | After 1 week, After 1 month, After 3 months
  Lipoatrrophy occurring after subcutaneous insulin injection will be determined by inspection and palpation.
lipohypertrophy | After 1 week, After 1 month, After 3 months
  lipohypertrophy occurring after subcutaneous insulin injection will be determined by inspection and palpation.
pain | during the first week, 1st month and the last week before the 3rd month
  Pain occurring after subcutaneous injection will be measured with "visual analog scale". These values will be written into the chart.
blood glucose level | during the first week, 1st month and the last week before the 3rd month
  Blood glucose values will be measured by patients with a blood glucose meter. These values will be written into the chart.

CONTACTS AND LOCATIONS:
Overall Officials: Azzet YÜKSEL, Principal Investigator — Kocaeli Sağlık ve Teknoloji Üniversitesi

IPD SHARING:
Plan to Share IPD: No